CLINICAL TRIAL: NCT06543784
Title: The New Wave of Preconception Carrier Screening: the Nurse Practitioner in the Lead?
Brief Title: Preconception Carrier Screening at the Erasmus MC
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Judith P.H. Robbemont, Nurse practitioner in training, Investigator, Erasmus Medical Center
Other Study IDs: 12716
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Inherited Genetic Conditions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Experts of experience: Health care professionals involved in preconception carrier screening at Amsterdam UMC, UMC Groningen and Australia
- Gynaecologists (in training)
- Midwives
- General practitioners
- Nurse practitioners and/or clinical geneticists
- Potential prospective patients who might want to undergo preconception carrier screening

SUMMARY:
Rationale A recent advisory report by the 'Health Council' has recommended that all prospective parents should have the opportunity to undergo preconception carrier screening. Consequently,there will no longer be any prerequisites for referring a couple. It is expected that there will be an increase in the number of prospective parents seeking counseling for preconception carrier screening. This is anticipated to result in an increase in the number of referrals, leading to several points of attention.

Objective(s) The aim of the research is to gather insights, perspectives, and experiences from healthcare professionals and prospective parents in order to design a care pathway for offering preconception carrier screening at Erasmus MC and the Rotterdam region. This will also include examining the role that nurse practitioners can play in this offering.

DETAILED DESCRIPTION:
Study type Exploratory research. Study population Healthcare professionals involved in preconception carrier screening and potential prospective parents who might want to undergo preconception carrier screening in the future. Methods Semi-structured interviews and focus groups will be used to explore topics which will be audio recorded and transcribed verbatim. The results will be analyzed by two to three researchers independently following the principles of grounded theory.

Burden and risks There are no risks associated with this research. For the interviewees and participants of the focus groups there is the burden of time investment. Recruitment and consent Health care professionals and potential prospective parents will be asked for participation in the study by the treating physician. If they consent to be approached, they will be informed about the study and contacted by the researcher. If willing to participate, an appointment for the interview/focus group is scheduled. Before the start of the interview/focus group, signed informed consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Health care professionals working with potential prospective parents.
* Potential prospective parents who might want to undergo preconception carrier screening in the future.

Exclusion Criteria:

* (Dutch) language proficiency not sufficient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care professionals involved in preconception carrier screening at Amsterdam UMC and UMC Groningen. Gynaecologists (in training), midwives, general practitioners, nurse practitioners and clinical geneticists from the clinical genetics department Erasmus MC and potential prospective parents who might want to undergo preconception carrier screening in the future.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Creating a pathway for preconception carrier screening using focus groups and interviews. | 1 year
  Using focus groups and interviews to gather insights, perspectives, and experiences from healthcare professionals and prospective parents in order to design a care pathway for offering preconception carrier screening at Erasmus MC and the Rotterdam region.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided